CLINICAL TRIAL: NCT04107181
Title: A Pilot Study Continuation to Assess the Use of an Introducer "Calla" During Cervical Cancer Screening
Brief Title: Pilot Study for Speculum Free Cervical Cancer Screening
Acronym: Calla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Korle-Bu Teaching Hospital, Accra, Ghana (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro00008173_1; R01CA239268-04 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: Pap smear
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Patient surveillance (Experimental): The introducer will be used during annual Pap smears for cervical cancer screening.
  Interventions: Device: Introducer "calla" device
- Healthy Volunteers (Experimental): There will be 2 types of healthy volunteers recruited to participate in this arm. The home study is to determine ease of use/feasibility of the introducer. The other group of healthy volunteers will be interviewed only. The goal of this study is to better understand how to improve women's health through learning about women's perceptions of their reproductive anatomy, specifically the cervix, comfort in discussing reproductive health topics with providers, and thoughts on two tools used to see the cervix.
  Interventions: Behavioral: Interviews only

INTERVENTIONS:
Device: Introducer "calla" device — The research introducer will be used after the patient consents prior to the annual pap smear.
  Arms: Patient surveillance
Behavioral: Interviews only — Healthy volunteer interviews
  Arms: Healthy Volunteers

SUMMARY:
The objective of the work described in this protocol is to determine the optical signatures of cervical dysplasia using optical technologies.

DETAILED DESCRIPTION:
This project is to assess if the introducer, "calla", can be used in place of a speculum during a routine Pap smear. For the patient arm, the introducer will be used in conjunction with standard of care procedures. The healthy volunteer arm will include taking the introducer home for a week to determine if each person can find their cervix without the help of a physician. As well as completing surveys on ease of use and demographics related to their medial history.

ELIGIBILITY:
Inclusion Criteria:

Healthy female

* Aged 21-65 years
* Have had a pelvic exam
* Have conversational proficiency in English
* Highest level of education attained

Exclusion Criteria:

- Pregnant women

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 305 (Estimated)
Dates: Start 2016-04-14 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of introducer | Up to 1 week (at time of pap smear for patients and up to 1 week for healthy volunteers)
  We will conduct interviews/surveys to determine if subjects enrolled prefer introducer over SOC speculum

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, PhD, Principal Investigator — Duke
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No